CLINICAL TRIAL: NCT05602012
Title: The Effect of Mindfulness Based Cognitive Counseling Group for Social Anxiety, Assertiveness and Self-Confidence in Nursing Students
Brief Title: Mindfulness Based Cognitive Counseling on Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Feride Ercan, Research Assistant, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FErcan
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Social Anxiety; Assertiveness; Self Confidence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Counseling (Experimental): The intervention was conducted in two groups with 25 participants/12-13 for each groups and two researchers per group. The program which consisted of eight sessions in total, was held once a week and each session lasted approximately 90-120 minutes.
  Interventions: Behavioral: Mindfulness based cognitive counseling group
- No Intervention (No Intervention): Participants will not be given an intervention until after they have completed the study. Data collection tools were applied to the students simultaneously with the intervention group, and after the follow-up test of the intervention group, a single-session information meeting will be held by the researchers for the students in the control group.

INTERVENTIONS:
Behavioral: Mindfulness based cognitive counseling group — Intervention: The sessions were conducted by the researchers who received training in the field of Mindfulness Based Cognitive Therapy. Sessions are structured as follows; 'Awareness and autopilot, living in our minds, tidying up the dispersed mind, recognizing the unpleasant/version, allowing, ways to take care of oneself, turning to face difficulties, being stuck in the past, living in the present?'
  Arms: Mindfulness Based Cognitive Counseling

SUMMARY:
The aim of the study is to determine the effect of group mindfulness based cognitive counseling on social anxiety, assertiveness and self-confidence in nursing students and the relationship of these variables to change over time.

DETAILED DESCRIPTION:
This is a randomized controlled and single-center study. The universe of the research consisted of nursing students who applied for counseling within the scope of the announcement made on the department web page. The research will be carried out in a state university, Faculty of Health Sciences, Department of Nursing between February 22, 2022 - December 23, 2022. In the study, the assignment of students to the intervention and control groups was made by simple randomization. Participant Information Form, Liebowitz Social Anxiety Scale, Self-Confidence Scale and Assertiveness Inventory will be used to collect the data of the study. Data collection tools will be applied three times simultaneously with the control group as a pre-test at the beginning of the study, as a post-test at the last session of the intervention group ( 2 month), and as a follow-up test 6 months after the last session of the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Liebowitz social anxiety scale score >50
* 18 years of age or older
* Volunteering to participate in the study

Exclusion Criteria:

* Diagnosed with a mental disorders
* History of participating in a counseling program
* Currently receiving individual or group counseling
* Unable to attend more than two sessions
* Diagnosed with a physical or mental disorder during group sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | Change from baseline to week 8 (2-month) and 6-month follow up
  A 24-item self-report measure that assesses fear and avoidance of social performance and social situations. The total scale score ranges from a minimum of 48 to a maximum of 192. An increase in the score indicates that the level of social anxiety and avoidance behavior are intensified.

SECONDARY OUTCOMES:
Assertiveness Inventory | Change from baseline to week 8 (2-month) and 6-month follow-up
  A 28-item self report inventory that assesses level of assertiveness. The total score that can be obtained from the scale is between a minimum of 28 and a maximum of 168. As the individual's score from the scale increases, the level of confidence increases.
Self Confidence Scale | Change from baseline to week 8 (2-month) and 6-month follow-up
  A 33-item self report scale that assesses level of self confidence. The highest score that can be obtained from the scale is 165 and the lowest score is 33. A high score from the scale indicates a high level of self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Feride Ercan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers will be able to reaad detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on the this PRS page.

REFERENCES:
- [Background] Demir S, Ercan F. The effectiveness of cognitive behavioral therapy-based group counseling on depressive symptomatology, anxiety levels, automatic thoughts, and coping ways Turkish nursing students: A randomized controlled trial. Perspect Psychiatr Care. 2022 Oct;58(4):2394-2406. doi: 10.1111/ppc.13073. Epub 2022 Mar 24. PMID 35332542